CLINICAL TRIAL: NCT03360747
Title: A Phase 2 Open-Label Study to Assess the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of AKCEA-ANGPTL3-LRx (ISIS 703802) Administered Subcutaneously to Patients With Familial Chylomicronemia Syndrome (FCS)
Brief Title: Phase 2 Study of AKCEA-ANGPTL3-LRx (ISIS 703802) in Participants With Familial Chylomicronemia Syndrome (FCS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 703802-CS3
Record Dates: First submitted 2017-11-18; First posted 2017-12-04 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Familial Chylomicronemia Syndrome; Lipoprotein Lipase Deficiency; Hyperlipoproteinemia Type 1
Keywords: Familial Lipoprotein Lipase Deficiency; Hyperlipoproteinemias; Familial Hyperlipoproteinemia Type 1; Hyperlipoproteinemia Type I; Hyperchylomicronemia, Familial; Lipoprotein Lipase Deficiency, Familial; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Lipid Metabolism, Inborn Errors; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome; Hyperlipoproteinemia Type I; Hyperlipoproteinemias; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Lipid Metabolism, Inborn Errors; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn | interventions — IONIS-ANGPTL3-LRx; vupanorsen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AKCEA-ANGPTL3-LRx 20 mg (Experimental): Participants received a subcutaneous (SC) injection of AKCEA-ANGPTL3-LRx, 20 milligrams (mg), weekly (QW) for 13-weeks of treatment period. Participants were followed up to Week 26.
  Interventions: Drug: AKCEA-ANGPTL3-LRx

INTERVENTIONS:
Drug: AKCEA-ANGPTL3-LRx — AKCEA-ANGPTL3-LRx at dose 20 mg, administered via SC injection QW.
  Other Names: ISIS 703802; IONIS-ANGPTL3-LRx; Vupanorsen

SUMMARY:
This is a single center, open-label study to evaluate the efficacy of AKCEA-ANGPTL3-LRx for reduction of triglyceride (TG) levels in participants with FCS.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetically confirmed chylomicronemia syndrome.
* Fasting triglycerides greater than or equal to (>=) 750 milligrams per deciliter (mg/dL) [8.4 millimoles per liter (mmol/L)] at Screening.

Key Exclusion Criteria:

* Diabetes mellitus if newly diagnosed or if glycated hemoglobin (HbA1c) >= 9.0%.
* Active pancreatitis within 2 weeks of screening.
* Acute coronary syndrome within 6 months of screening.
* Major surgery within 3 months of screening.
* Treatment with Glybera therapy within 2 years of screening.
* Previous treatment with AKCEA-ANGPTL3-LRx.
* Have any other conditions in the opinion of the investigator which could interfere with the patient participating in or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigative Site, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 study site in Canada from 21-December-2017 to 4-September-2018.
Pre-assignment Details: A total of 4 participants were screened, 3 of whom were enrolled and treated with at least one dose of study drug and were included in the analysis. This study consisted of up to an 8-week screening period, a 13-week treatment period and a 13-week follow-up (post-treatment evaluation) period.
Period: Overall Study
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Started | 3
Completed | 2
Not Completed | 1
Not completed — Voluntary Withdrawal | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- AKCEA-ANGPTL3-LRx 20 mg: Participants received a SC injection of AKCEA-ANGPTL3-LRx, 20 mg, QW for 13-weeks of treatment period. Participants were followed up to Week 26.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (15.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Fasting Triglycerides (TG) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 2299.50 (961.139)
Fasting Angiopoietin-Like 3 (ANGPTL3) [Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)] | 62.433 (8.9030)
Fasting Total Cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 316.50 (81.957)
Fasting Non-High Density Lipoprotein Cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 301.17 (82.791)
Fasting Apolipoprotein B (ApoB) [Mean (Standard Deviation); unit: mg/dL] | 72.65 (9.406)
Fasting High Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 15.3 (1.15)
Fasting Apolipoprotein A-1 (ApoA-1) [Mean (Standard Deviation); unit: mg/dL] | 94.7 (7.51)
Fasting Very Low Density Lipoprotein Cholesterol (VLDL-C) [Mean (Standard Deviation); unit: mg/dL] | 272.67 (89.326)
Fasting Low Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 28.50 (6.946)
Maximum Postprandial Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 2454.81 (1019.963)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Month 3 in Fasting Triglycerides (TG)
Description: Baseline was defined as the average of Day 1 predose fasting assessment and the last fasting measurement prior to Day 1 pre-dose fasting assessment. Month 3 was defined as the average of Week 13 and Week 14 fasting assessments.
Time Frame: Baseline to Month 3
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
mg/dL | -550.00 (431.471)

2. Primary Outcome: Percent Change From Baseline to Month 3 in Fasting Triglycerides (TG)
Description: as for outcome 1
Time Frame: Baseline to Month 3
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
percent change | -32.83 (31.994)

3. Secondary Outcome: Absolute Change From Baseline to Month 3 in Fasting Angiopoietin-Like 3 (ANGPTL3)
Description: as for outcome 1
Time Frame: Baseline to Month 3
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
ng/mL | -31.983 (5.4773)

4. Secondary Outcome: Percent Change From Baseline to Month 3 in Fasting Angiopoietin-like 3 (ANGPTL3)
Description: as for outcome 1
Time Frame: Baseline to Month 3
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
percent change | -51.249 (4.9093)

5. Secondary Outcome: Fasting Lipid and Lipoprotein Measurements at Month 3
Description: Fasting lipid and lipoprotein measurements included non-HDL-C, ApoB, HDL-C, ApoA-1, VLDL-C and LDL-C. Month 3 was defined as the average of Week 13 and Week 14 fasting assessments.
Time Frame: Month 3
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
mg/dL
  Non-HDL-C | 217.33 (119.618)
  ApoB | 64.53 (4.899)
  HDL-C | 13.0 (1.00)
  ApoA-1 | 77.3 (6.03)
  VLDL-C | 190.17 (128.861)
  LDL-C | 27.17 (10.324)

6. Secondary Outcome: Absolute Change From Baseline to Month 3 in Other Fasting Lipid Parameters
Description: Other fasting lipid measurements included total cholesterol (TC), non-HDL-C, ApoB, HDL-C, ApoA-1, VLDL-C, and LDL-C. Baseline was defined as average of Day 1 predose fasting assessment and last fasting measurement prior to Day 1 pre-dose fasting assessment. Month 3 was defined as the average of Week 13 and Week 14 fasting assessments.
Time Frame: Baseline to Month 3
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
mg/dL
  Absolute Change From Baseline to Month 3 in TC | -86.17 (48.581)
  Absolute Change From Baseline to Month 3:Non-HDL-C | -83.83 (48.235)
  Absolute Change From Baseline to Month 3 in ApoB | -8.12 (5.352)
  Absolute Change From Baseline to Month 3 in HDL-C | -2.3 (0.58)
  Absolute Change From Baseline to Month 3 in ApoA-1 | -17.3 (11.93)
  Absolute Change From Baseline to Month 3 in VLDL-C | -82.50 (51.215)
  Absolute Change From Baseline to Month 3 in LDL-C | -1.33 (3.753)

7. Secondary Outcome: Percent (%) Change From Baseline to Month 3 in Other Fasting Lipid Parameters
Description: Other fasting lipid measurements included TC, non-HDL-C, ApoB, HDL-C, ApoA-1, VLDL-C, and LDL-C. Baseline was defined as average of Day 1 predose fasting assessment and last fasting measurement prior to Day 1 pre-dose fasting assessment. Month 3 was defined as the average of Week 13 and Week 14 fasting assessments.
Time Frame: Baseline to Month 3
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
percent change
  % Change From Baseline to Month 3 in TC | -30.39 (20.436)
  % Change From Baseline to Month 3 in Non-HDL-C | -31.49 (21.832)
  % Change From Baseline to Month 3 in ApoB | -10.73 (6.021)
  % Change From Baseline to Month 3 in HDL-C | -15.2 (3.22)
  % Change From Baseline to Month 3 in ApoA-1 | -17.8 (10.97)
  % Change From Baseline to Month 3 in VLDL-C | -36.03 (28.044)
  % Change From Baseline to Month 3 in LDL-C | -6.47 (13.426)

8. Secondary Outcome: Change From Baseline to Day 92 in Maximum Postprandial Triglycerides (TG)
Description: Participants consumed standardized pre-cooked meals (lunches and dinners and instructions for breakfasts and snacks) for 2 days prior to the postprandial assessments. Change from Baseline to Day 92 in maximum postprandial TG was assessed.
Time Frame: Baseline to Day 92
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 2
mg/dL | -338.0 (38.22)

9. Secondary Outcome: Number of Participants Who Experienced Abdominal Pain During the Treatment Period
Time Frame: Days 1, 29, 57 and 92
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
Participants | 1

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product. A TEAE was defined as any AE starting on or after the first dose of the study drug.
Time Frame: From time of informed consent to end of follow-up period (Up to Week 26)
Population: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: From time of informed consent to end of follow-up period (Up to Week 26).
Description: Safety set included all participants who were enrolled and received at least 1 dose of study drug.
Arm/Group | AKCEA-ANGPTL3-LRx 20 mg
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKCEA-ANGPTL3-LRx 20 mg (N=3)
Asthenia (General disorders) | 1
Influenza like illness (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Vertigo positional (Ear and labyrinth disorders) | 1
Influenza (Infections and infestations) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Loss of libido (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT03360747/Prot_SAP_000.pdf